CLINICAL TRIAL: NCT04030624
Title: Remote Electronic Patient Monitoring in Gastrointestinal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding discontinued due to changes in corporate structures
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph A. Greer, Ph.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-329
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Remote Electronic Patient Monitoring (Experimental): * The Remote Electronic Patient Monitoring intervention will entail monitoring of vital sign data and patient reported assessments to address and manage any concerning issues identified.
  * The Remote Patient Monitoring system uses algorithms that can indicate when patient vitals and patient-reported outcomes have changed.
  * Automatic patient surveys are sent to the patient with results displayed on the clinician user interface (i.e., dashboard) on a computer located in the clinical area.
  * Qualitative interviews with patient participants and their oncology clinicians using a semi-structured interview guide will be conducted.
  Interventions: Device: Remote Electronic Patient Monitoring

INTERVENTIONS:
Device: Remote Electronic Patient Monitoring — The Remote Patient Monitoring intervention is a remote monitoring system intended for use by healthcare professionals for the collection of physiological data in home and healthcare settings. Patient information is displayed on a computer located at the medical institution. Throughout the day, patient data from the remote monitoring system are presented on the clinician user interface (e.g., temperature, blood pressure, heart rate, respiration rate). Data are transmitted from sensors to the patient's smart phone.

SUMMARY:
The goal of this research study is to evaluate a program that involves remote electronic monitoring of vital signs and symptoms of patients with gastrointestinal cancer who were recently hospitalized at Massachusetts General Hospital or presented to the oncology clinic for an unplanned, urgent visit.

DETAILED DESCRIPTION:
Patients with gastrointestinal cancer often experience troublesome symptoms and side effects related to the cancer and its treatment. Unfortunately, patients commonly require hospital admission or urgent clinic visits to help manage uncontrolled symptoms. For this study, the investigators seek to determine if a program that entails remote electronic monitoring may improve the overall care experience of patients with gastrointestinal cancer who have urgent care needs.

The investigators are asking the participants to take part in this research study because the participants are currently hospitalized at Massachusetts General Hospital or recently presented to the oncology clinic for an urgent visit, and are receiving treatment at the Cancer Center. The goal of this study is to test a program that involves remote electronic monitoring of vital signs and patient-reported health outcomes. This study is a pilot study, and the investigators are evaluating the feasibility of delivering the program, the acceptability and satisfaction with the program, changes in the quality of life and symptoms of patients who receive the program, as well as the frequency of urgent hospital visits while the patient is in the program.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosed with gastrointestinal cancer
* Hospitalized at Massachusetts General Hospital (MGH) or presenting to the ambulatory MGH oncology clinic for an unplanned, urgent visit
* Planning to receive outpatient care at the MGH Cancer Center
* Ability to read and respond to questions in English

Exclusion Criteria:

* Uncontrolled psychiatric illness or impaired cognition that would interfere with completing study procedures
* Enrolled in hospice
* Planning to be discharged to any location other than their home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
The Feasibility of Remote Electronic Patient Monitoring Intervention | 4 weeks
  The intervention will be deemed feasible if at least 50% (95% confidence interval +/- 13%) of patients agree to participate in the study and sign informed consent, and if participants wear the Remote Electronic Patient Monitoring device ≥ 50% (95% confidence interval +/- 13%) of the time within the two weeks following the baseline time point.

SECONDARY OUTCOMES:
Proportion of participants completing self-reported symptom monitoring through the remote electronic monitoring device during study period | 4 weeks
Proportion of participants completing vital sign monitoring through the remote electronic monitoring device during study period | 4 weeks
Number of concerning issues identified per patient during study period | 4 weeks
Number of intervention-triggered phone calls from clinicians required per patient as well as average duration of these calls during study period | 4 weeks
Number of intervention-triggered emails generated to the primary oncology team during study period | 4 weeks
Proportion of intervention-triggered events that are not clinically acted upon (i.e., no change in patient care based on an intervention trigger) during study period | 4 weeks
Acceptability of Remote Electronic Patient Monitoring Intervention | 4 weeks
  Participant report of perceptions of the usefulness, effectiveness, and relevance of the intervention per acceptability ratings and qualitative interviews with patient participants and their clinicians.
Patient-Reported Quality of Life | 2 weeks and 4 weeks
  Change in patient-reported quality of life from baseline to 2 and 4 weeks per the Functional Assessment of Cancer Therapy-General
Patient-Reported Symptoms | 2 weeks and 4 weeks
  Change in patient-reported symptoms from baseline to 2 and 4 weeks per the Edmonton Symptom Assessment System-revised
Patient-Reported Depression and Anxiety Symptoms | 2 weeks and 4 weeks
  Change in patient-reported depression and anxiety symptoms from baseline to 2 and 4 weeks per the Patient Health Questionnaire-4
Health Care Utilization | 4 weeks
  Number of urgent clinic visits, emergency department visits, and hospital admissions during study period

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Greer, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation